CLINICAL TRIAL: NCT04037046
Title: Clinical Trial to Evaluate the Acceptance and Viability of Three Strategies in Birth Cohort Hepatitis C Screening
Brief Title: Integrating Hepatitis C Screening With Dried Blood Spot Testing Into Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Manuel Hernandez-Guerra, MD, Principal Investigator, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DBS_FOT
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Screening HCV with DBS at primary care centers (Experimental): Patients assigned to the strategy 1 will receive an invitation letter for HCV screening with DBS at the primary care center to be performed by the general practitioner
  Interventions: Behavioral: Screening HCV at primary care center
- Screening HCV and CCR with FOT at primary care centers (Active Comparator): Patients assigned to the strategy 2 will receive an invitation letter for HCV screening with DBS and CCR screening with FOT at the primary care center to be performed by the general practitioner
  Interventions: Behavioral: Screening HCV attached onto CCR screening
- Self-testing at home for screening HCV and CCR (Active Comparator): Patients assigned to the strategy 3 will receive an invitation letter for self-testing at home for HCV screening with DBS, and CCR screening with FOT
  Interventions: Behavioral: Screening HCV attached onto CCR screening by self-testing

INTERVENTIONS:
Behavioral: Screening HCV attached onto CCR screening — Patients assigned to this strategy will receive an invitation letter for HCV screening with DBS and CCR screening with FOT at the primary care center to be performed by the general practitioner
  Arms: Screening HCV and CCR with FOT at primary care centers
Behavioral: Screening HCV attached onto CCR screening by self-testing — Patients assigned to this strategy will receive an invitation letter for self-testing for HCV screening with DBS, and CCR screening with FOT
  Arms: Self-testing at home for screening HCV and CCR
Behavioral: Screening HCV at primary care center — DBS for HCV screening at primary care center
  Arms: Screening HCV with DBS at primary care centers

SUMMARY:
The main purpose of the study is to compare the acceptance and viability of three strategies aimed to screen hepatitis C virus (HCV) infection in a birth cohort by: a) invitation letter offering HCV screening with dried blood spot (DBS) testing at the primary care center, b) invitation letter offering both HCV and colorectal cancer (CCR) screening with faecal occult test (FOT) at the primary care center, and c) invitation letter offering self-collected screening at home for HCV and CCR.

DETAILED DESCRIPTION:
This is a prospective, randomized, study in which subjects of four different health areas will be invited to participate in three different screening strategies for HCV.

Hepatologists from a tertiary care hospital and general practitioners from four health areas will participate coordinating the study, to first select potential candidates for the study (subjects between 50 and 70 years old of the four areas) and secondly, randomize and include 150 subjects of each area into the three strategies (50 subjects each). The strategies include offering by letter screening at the local primary care center for HCV by using dried blood spot (DBS) testing, screening for HCV and colorectal cancer (CCR) using faecal occult test (FOT) at the primary care center, and self-testing at home-collection with DBS and FOT to be performed by the subject and sent by postal office. Subjects will receive an invitation and informative letter and will be ask to sign the informed consent to participate.

In all the planned strategies subjects will be asked to complete a questionnaire that includes demographic variables. After two months of sending the letters without response, researchers will contact subjects by phone to complete a survey to confirm they received the letter and asking for factors of non-participation.

The hypothesis of the study is that subjects in the risk of having HCV are willing to be screened for HCV infection if offered and that the acceptance will be improved if attached to CCR screening and even higher if the tests are offered to be self-screened.

For the present study, a 15% improvement in the participation (acceptance of the screening strategy) was hypothesized in the group of patients receiving the strategy 2 (and 3) compared to the strategy 1. Taking into account a power of 80%, alpha error of 5% and losses of 20% will require 200 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-70 years
* Subjects attending selected primary care centers
* Willing to participate (informed consent signed)

Exclusion Criteria:

-

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Acceptance of the interventions | 12 months
  overall screening rate (number of subjects participating after enrollment)

SECONDARY OUTCOMES:
Feasibility of the intervention measuring quality of spotted cards | 12 months
  the validity of specimens (defined as enough blood sample to fill at least one spot in the card) of DBS tests performed at primary care centers and by self-testing at home
Subject characteristics associated with participation and feasibility of the different strategies | 12 months
  Demographic characteristics associated with participation and feasibility of the different strategies
Effectiveness of each strategy: rate of HCV positivity | 12 months
  rate of HCV positivity

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hernandez-Guerra, MD, Principal Investigator — MD
Locations (1):
- Manuel Hernandez-Guerra, MD, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buti M, Dominguez-Hernandez R, Casado MA, Sabater E, Esteban R. Healthcare value of implementing hepatitis C screening in the adult general population in Spain. PLoS One. 2018 Nov 28;13(11):e0208036. doi: 10.1371/journal.pone.0208036. eCollection 2018. PMID 30485377
- [Background] Zuure FR, Urbanus AT, Langendam MW, Helsper CW, van den Berg CH, Davidovich U, Prins M. Outcomes of hepatitis C screening programs targeted at risk groups hidden in the general population: a systematic review. BMC Public Health. 2014 Jan 22;14:66. doi: 10.1186/1471-2458-14-66. PMID 24450797
- [Background] Tuaillon E, Mondain AM, Meroueh F, Ottomani L, Picot MC, Nagot N, Van de Perre P, Ducos J. Dried blood spot for hepatitis C virus serology and molecular testing. Hepatology. 2010 Mar;51(3):752-8. doi: 10.1002/hep.23407. PMID 20043287